CLINICAL TRIAL: NCT00609011
Title: Dose Finding Phase 1 Study of the Treatment of Metastatic Melanoma With MPC-6827 in Combination With Temozolomide
Brief Title: Phase 1 Study of MPC-6827 and Temozolomide in Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Andrew P. Beelen, MD / Sr. Director of Clinical Research, Myriad Pharmaceuticals
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPC-6827-07-005
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2010-08-23 (Estimated); Status verified 2010-08

CONDITIONS: Metastatic Melanoma
Keywords: Melanoma; Metastatic
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis | interventions — verubulin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MPC-6827 + Temozolomide — MPC-6827 at 2.1mg/m2, 2.7mg/m2 or 3.3mg/m2 administered by intravenous infusion over 2 hours once weekly for three weeks in a 4 week cycle. Temozolomide at 85 mg/m2 administered orally daily for 21 days in a 4 week cycle.

SUMMARY:
This is an open-label, dose finding, multiple-dose study in subjects with metastatic melanoma. Three dose levels of MPC-6827 will be administered with temozolomide to three separate cohorts. Study endpoints will include determination of the maximum tolerated dose, determination of dose limiting toxicities, and evaluation of evidence of anti-tumor activity of MPC-6827 when given with temozolomide.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven melanoma
* For subjects with brain metastases that require radiation, therapy must have been completed at least 4 weeks prior to Day 1 of Study Drug
* Have unresectable melanoma with measurable metastases
* Be a minimum of 4 weeks since prior surgical resection or major surgical procedure and a minimum of 2 weeks since chemotherapy/ biochemotherapy
* Performance score of Karnofsky ≥ 60%, or Eastern Cooperative Oncology Group (ECOG) ≤ 2, or WHO ≤ 2
* If steroids are needed, be on a stable or decreasing dose of steroids for at least 1 week

Exclusion Criteria:

* Hypersensitivity to Cremophor EL
* Have current/active intratumor hemorrhage by CT/MRI within 3 weeks prior to Day 1 of Study Drug confirmed by CT/MRI
* Have ocular melanoma
* Have primary intradural melanoma or leptomeningeal involvement
* Have cardiovascular disease (unstable angina or MI)
* Have cerebrovascular disease (stroke and/or TIA)
* Have uncontrolled hypertension
* Have a cardiac ejection fraction < 50%
* Have Troponin-I elevated above the normal range

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2008-03; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability; Maximum Tolerated Dose | After each cohort is enrolled

SECONDARY OUTCOMES:
Pharmacokinetics | Cycle 1
Antitumor Activity | Screening, end of each cycle, end of study

CONTACTS AND LOCATIONS:
Overall Officials: Andrew P. Beelen, MD, Study Director — Myrexis Inc.
Locations (5):
- United States (5):
  - The Angeles Clinic, Los Angeles, California
  - Cancer Centers of Florida, Ocoee, Florida
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute at the University of Utah, Salt Lake City, Utah